CLINICAL TRIAL: NCT04112407
Title: The Effect of Pretreatment for Propionibacterium Acnes on Surgical Site Burden in Shoulder Arthroplasty; a Pilot Study
Brief Title: The Effect of Pretreatment for Propionibacterium Acnes on Surgical Site Burden in Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Joseph Zimmerman, MD, Attending Orthopaedic Surgeon, Department of Surgery, Division of Orthopaedic Surgery,, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5316
Record Dates: First submitted 2019-07-22; First posted 2019-10-02 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Shoulder Arthroplasty
Keywords: P. Acnes; shoulder arthroplasty; blue light therapy; benzoyl peroxide
MeSH Terms: interventions — Phototherapy; Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control (Experimental): Standard preparation of the surgical site without P. acnes pretreatment
  Interventions: Other: Control
- BPO Group (Experimental): Pretreatment with 10% Benzoyl peroxide body wash for two consecutive days of washes prior to surgery at home. The anterior shoulder area is wet before treatment; the wash is massaged in for 20 seconds producing a lather and washed off, patting dry.
  Interventions: Drug: Benzyl Peroxide
- BPO and Phototherapy (Experimental): 2 days of benzoyl peroxide washes and 3 treatments of blue light phototherapy. Pretreatment with 10% Benzoyl peroxide body wash for two consecutive days of washes prior to surgery at home. The anterior shoulder area is wet before treatment; the wash is massaged in for 20 seconds producing a lather and washed off, patting dry. The blue light phototherapy is administered to the shoulder for 3 minutes on three occasions; 2 days before, the day before surgery and in the preoperative area by the patient.
  Interventions: Device: Blue Light Phototherapy; Drug: Benzyl Peroxide

INTERVENTIONS:
Device: Blue Light Phototherapy — Phototherapy in the blue light spectrum
  Other Names: Phototherapy
  Arms: BPO and Phototherapy
Drug: Benzyl Peroxide — Benzyl peroxide wash to be used preoperatively during showering to the operative shoulder site.
  Other Names: BPO
  Arms: BPO Group; BPO and Phototherapy
Other: Control — Standard surgical site preparation with no P. acnes pretreatment
  Arms: Control

SUMMARY:
Cutibacterium acnes - formally known as Propionibacter acnes (P. acnes) is the most common pathogen associated with prosthetic joint infection of the shoulder. Despite current skin preparation techniques, P. acnes is encountered at the skin surface and at the natural reservoir in the sebaceous glands during the surgical exposure; current levels of exposure are implicated in overall prosthetic infection risk. Therefore, this study endeavors to decrease P. acnes burden at the surgical incision using preoperative blue light phototherapy and benzyl peroxide washes targeting both the skin surface and sebaceous glands.

DETAILED DESCRIPTION:
The study hypotheses will be tested using a prospective randomized-controlled trial of the effect of combination blue spectrum phototherapy and benzoyl peroxide on P. acnes at the shoulder arthroplasty surgical site. Accordingly, it will conform to the CONSORT (Consolidated Standards of Reporting Trials) guidelines. Subjects presenting to our Orthopaedic department will be randomized to one of three study arms:

1. Control: standard preparation of the surgical site without P. acnes pretreatment
2. BPO group: Pretreatment with 2 days of washes prior to surgery
3. BPO and Phototherapy: 2 days of washes with 3 treatments of blue spectrum phototherapy

Patients will be seen at our office will be consented and recruited into the study. Subjects will have standard of care evaluation including: radiographs, preoperative labs and clearances. If selected and agreeable, treatment with phototherapy will involve the application of three sessions lasting 3 minutes preoperatively; the sessions will be conducted by the patient at home for two days prior to surgery and in the preoperative holding area. During each application, protective eyewear will be used. For patients in the BPO groups, a 10% benzoyl peroxide wash will be used globally on the operative shoulder and axilla during showering. An educational leaflet will outline the surgical field in addition to temporary demarcation at the time of BPO pickup at the office. Additional tests, imaging or procedures will be at the discretion of the treating physician and documented during the study. During the postoperative visit at 10-14 days, the post operative wound will be assessed in the standard manner. Final culture results will be recorded for each patient and documented in the study database.

* The surgical site will be prepared in usual fashion with Chloroprep and the patients will receive preoperative Cefazolin (or vancomycin based on penicillin allergy)
* Following both draping and skin incision, the surgeons gloves will be changed; any blades used in the skin incision will also be discarded
* Intraoperative cultures will be taken following established protocols, published in the literature: an excisional biopsy 1cm long and 3mm wide will be taken from the medial wound edge at the time of incision; the superficial dermal tissue will be swabbed immediately after the biopsy is taken and finally, a swab of the glenohumeral (shoulder) joint will be performed prior to closure at the end of the procedure and after insertion of the implant.
* Specimens will be transported to the laboratory adjoining the operating room at our institution within 1 hour of harvesting and processed by microbiology technicians in a laminar flow biological safety hood. Tissue from the skin edge will be homogenized in sterile saline solution and plated on media: blood agar, chocolate agar, Brucella agar, MacConkey agar, Columbia nalidixic acid agar and phenylethyl alcohol anaerobic blood agar. All media will be incubated at 37C for 14 days.
* Specimens will be incubated for 14 days in aerobic and anaerobic media to detect P acnes and other organisms
* Culture results will not be discussed with patients; patients will be consented to not know their results as they are not clinically significant
* Prophylactic antibiotic treatment of positive cultures will not be performed in any case.

ELIGIBILITY:
Inclusion Criteria

* All patients presenting to the practice that require a shoulder arthroplasty procedure
* English fluency and literacy
* Able to provide informed consent
* Older than 18 years of age
* Surgical indications including: primary arthritis, rotator cuff arthropathy, post-traumatic arthritis
* Primary total shoulder, hemiarthroplasty, primary reverse total shoulder or shoulder resurfacing

Exclusion Criteria

* Subjects who have had a prior infection of the affected shoulder joint
* Recent steroid injection to the shoulder in the past 6 months
* Previous open or arthroscopic procedure of the shoulder joint
* Recent antibiotic use (within 90 days)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of total culture positivity during shoulder arthroplasty | 14 days in culture
  To compare the rates of P. Acnes culture positivity (including all samples) between groups. Therein, assessing the efficacy of the interventions to decrease P. Acnes burden (measured by the rate of culture positivity) in surgical field.

SECONDARY OUTCOMES:
Correlation of the rate of superficial culture positivity and the rate deep culture positivity during shoulder arthroplasty | 14 days in culture
  To investigate the correlation between the rate of positive deep cultures in samples taken at the end of surgery (1 deep swab) and the rate of superficial culture positivity of samples taken at the beginning of the case (incisional biopsy and superficial dermal swab). It is theorized that P. Acnes in the superficial wound is propagated to the deeper tissues during surgery, impacting deep culture rates and possibly contributing to prosthetic joint infection risk.

CONTACTS AND LOCATIONS:
Overall Officials: Ian D Hutchinson, MD, Study Director — Albany Medical College
Locations (2):
- United States (2):
  - Albany Medical Center, Albany, New York
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frangiamore SJ, Saleh A, Grosso MJ, Alolabi B, Bauer TW, Iannotti JP, Ricchetti ET. Early Versus Late Culture Growth of Propionibacterium acnes in Revision Shoulder Arthroplasty. J Bone Joint Surg Am. 2015 Jul 15;97(14):1149-58. doi: 10.2106/JBJS.N.00881. PMID 26178890
- [Result] Pottinger P, Butler-Wu S, Neradilek MB, Merritt A, Bertelsen A, Jette JL, Warme WJ, Matsen FA 3rd. Prognostic factors for bacterial cultures positive for Propionibacterium acnes and other organisms in a large series of revision shoulder arthroplasties performed for stiffness, pain, or loosening. J Bone Joint Surg Am. 2012 Nov 21;94(22):2075-83. doi: 10.2106/JBJS.K.00861. PMID 23172325
- [Result] Saltzman MD, Nuber GW, Gryzlo SM, Marecek GS, Koh JL. Efficacy of surgical preparation solutions in shoulder surgery. J Bone Joint Surg Am. 2009 Aug;91(8):1949-53. doi: 10.2106/JBJS.H.00768. PMID 19651954
- [Result] Rao AJ, Chalmers PN, Cvetanovich GL, O'Brien MC, Newgren JM, Cole BJ, Verma NN, Nicholson GP, Romeo AA. Preoperative Doxycycline Does Not Reduce Propionibacterium acnes in Shoulder Arthroplasty. J Bone Joint Surg Am. 2018 Jun 6;100(11):958-964. doi: 10.2106/JBJS.17.00584. PMID 29870447
- [Result] Lee MJ, Pottinger PS, Butler-Wu S, Bumgarner RE, Russ SM, Matsen FA 3rd. Propionibacterium persists in the skin despite standard surgical preparation. J Bone Joint Surg Am. 2014 Sep 3;96(17):1447-50. doi: 10.2106/JBJS.M.01474. PMID 25187583
- [Result] Falconer TM, Baba M, Kruse LM, Dorrestijn O, Donaldson MJ, Smith MM, Figtree MC, Hudson BJ, Cass B, Young AA. Contamination of the Surgical Field with Propionibacterium acnes in Primary Shoulder Arthroplasty. J Bone Joint Surg Am. 2016 Oct 19;98(20):1722-1728. doi: 10.2106/JBJS.15.01133. PMID 27869623
- [Result] Canavan TN, Chen E, Elewski BE. Optimizing Non-Antibiotic Treatments for Patients with Acne: A Review. Dermatol Ther (Heidelb). 2016 Dec;6(4):555-578. doi: 10.1007/s13555-016-0138-1. Epub 2016 Aug 19. PMID 27541148
- [Result] Kolakowski L, Lai JK, Duvall GT, Jauregui JJ, Dubina AG, Jones DL, Williams KM, Hasan SA, Henn RF 3rd, Gilotra MN. Neer Award 2018: Benzoyl peroxide effectively decreases preoperative Cutibacterium acnes shoulder burden: a prospective randomized controlled trial. J Shoulder Elbow Surg. 2018 Sep;27(9):1539-1544. doi: 10.1016/j.jse.2018.06.012. Epub 2018 Jul 24. PMID 30054245
- [Result] Dai T, Gupta A, Murray CK, Vrahas MS, Tegos GP, Hamblin MR. Blue light for infectious diseases: Propionibacterium acnes, Helicobacter pylori, and beyond? Drug Resist Updat. 2012 Aug;15(4):223-36. doi: 10.1016/j.drup.2012.07.001. Epub 2012 Jul 28. PMID 22846406
- [Result] Kawada A, Aragane Y, Kameyama H, Sangen Y, Tezuka T. Acne phototherapy with a high-intensity, enhanced, narrow-band, blue light source: an open study and in vitro investigation. J Dermatol Sci. 2002 Nov;30(2):129-35. doi: 10.1016/s0923-1811(02)00068-3. PMID 12413768
- [Result] Ash C, Dubec M, Donne K, Bashford T. Effect of wavelength and beam width on penetration in light-tissue interaction using computational methods. Lasers Med Sci. 2017 Nov;32(8):1909-1918. doi: 10.1007/s10103-017-2317-4. Epub 2017 Sep 12. PMID 28900751
- [Result] Oplander C, Hidding S, Werners FB, Born M, Pallua N, Suschek CV. Effects of blue light irradiation on human dermal fibroblasts. J Photochem Photobiol B. 2011 May 3;103(2):118-25. doi: 10.1016/j.jphotobiol.2011.02.018. Epub 2011 Feb 26. PMID 21421326